CLINICAL TRIAL: NCT02396173
Title: Does the Knowledge of a "Non-return to Work" Predictive Score Influence Vocational Rehabilitation After Orthopaedic Trauma?
Brief Title: Does the Knowledge of a "Non-return to Work" Predictive Score Influence Vocational Rehabilitation?
Acronym: WORRK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Romande de Readaptation (Network)
Collaborators: University of Applied Sciences of Western Switzerland (Other)
Responsible Party: Principal Investigator, François Luthi, Senior lecturer and researcher, Clinique Romande de Readaptation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: CliniqueRR-03
Record Dates: First submitted 2015-03-10; First posted 2015-03-24 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Pain
Keywords: disability; vocational; rehabilitation; prediction
MeSH Terms: conditions — Pain | interventions — Risk Factors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risk Score for non-return to work (Experimental): The WORRK model is a predictive tool (19 items) of the non-return to work risk useful for all kinds of orthopaedic trauma and for patients needing vocational rehabilitation. It is constructed with variables independent of the patient's education and language fluency. It is a short patient's bedside tool and takes less than 20 minutes.
  Interventions: Other: Risk Score for non-return to work
- Control group (No Intervention): In this group the medical staff will not be informed about the risk score (WORRK).

INTERVENTIONS:
Other: Risk Score for non-return to work — The WORRK tool will be filled in for all patients, even the patients in the control group. However, the probability score will only be accessible for the medical doctors in the intervention group, along with guidelines for interpretation ("1. With a probability score over 50% (not to return to work), patient's allocation to the "Evaluation Pathway" should be considered" "2. With a probability score over 70% (not to return to work), the "Evaluation Pathway" is probably the most suitable choice").
  Arms: Risk Score for non-return to work

SUMMARY:
Background: Orthopaedic trauma are a leading cause of long-lasting sick-leave and persistent disability. People suffering from persistent sick-leave often need vocational rehabilitation (VR). Vocational programs are planned to improve the likelihood of returning to work (RTW). Physical conditioning, professional evaluation and training, as well as psychological and social interventions are the core of the treatments. Efficiency of these programs is moderate and there is scope for improvements. For instance, rehabilitation programs tailored to the individual needs and potentials are called for. However, the allocation remains difficult. Decision-supportive tools may be convenient to achieve this goal. Recently, the WORRK model was proposed to assess early on the risk of non-returning to work for those patients. The main goal of this research is to measure if the WORRK model improves patients' allocation to different vocational programs according to their "non-return to work" risk.

DETAILED DESCRIPTION:
Methods:

Vocational inpatients after orthopaedic trauma (n=280), aged between 18-60 years. Three different vocational pathways can be selected: Simple (for patients with low "non-return to work" risk, 5 weeks stay), Coaching (intermediate risk, 5 weeks), Evaluation (high risk, 3 weeks). Design: randomized-controlled trial. In the intervention group, the probability not to return to work estimated with the WORRK model will be offered to the clinician team before the allocation decisions. In the control group, the probability will also be estimated but not known by the clinician team. The primary outcome is the proportion of patients allocated to the Evaluation Pathway. Secondary outcomes: the patients' satisfaction is not worse in the intervention group; the decisions makers' satisfaction with the information available for the decision process is better in the intervention group; the proportion of patients changing the treatment pathway during the vocational stay is not higher in the intervention group; and the calibration of the WORRK model remains satisfactory; the non-return to work rate is not higher in the intervention group than in the control group (follow-up at 3, 12, and 24 months);

Relevance and impact:

The investigators expect that the WORRK model will improve the efficiency of vocational rehabilitation after orthopedic trauma. This will due to better allocation to the vocational pathways according to the patients' risk profile. If this is the case, an increase of the shorter vocational program is expected without jeopardizing the chance of returning to work and the patient satisfaction with quality of care. The ability of the WORRK model to detect patients with similar risk profiles could also strengthen the interest for this decision-supportive tool in clinical practice and trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for a vocational rehabilitation programme after an orthopaedic trauma

Exclusion Criteria:

* Severe traumatic brain injury at time of accident (Glasgow coma Scale ≤8)
* Spinal Cord Injury
* Not capable of judgment
* Under legal custody

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Allocation to the evaluation pathway (proportion of patients allocated to the Evaluation Pathway) | 10 months
  The primary outcome in the WORRK study is the proportion of patients allocated to the Evaluation Pathway.

SECONDARY OUTCOMES:
Return to work rate | 24 months
  The non-return to work rate will be assessed by questionnaire at 3, 12 and 24 months after discharge.
the patients' satisfaction is not worse in the intervention group | 10 months
  At discharge patients will fill a questionnaire to assess their satisfaction regarding the treatments received.
the decisions makers' satisfaction with the information available for the decision process is better in the intervention group | 10 months
  Medical staff will assess efficiency of the intervention through a questionnaire
the proportion of patients changing the treatment pathway during the vocational stay is not higher in the intervention group | 10 months
  To assess if patients change their clinical pathway during hospitalization. Is there any differences between the intervention and control groups.
the calibration of the WORRK model remains satisfactory | 24 months
  We will perform a new validation of the WORRK model on the population recruited from this study. The performance of the WORRK prediction tool will be assessed with measures for calibration and discrimination. For calibration we will plot the expected against the observed proportion of non-return to work per predicted risk group. Furthermore, we will use the Hosmer-Lemeshow test to define statistical significance of the calibration. For discrimination, we will plot the ROC-curve and calculate Areas under the ROC-curve (AUC). We consider the performance of the WORRL acceptable if there is good calibration (i.e. intercept not statistically different from 0 and slope of 1) and if the AUC is larger than 0.7.

CONTACTS AND LOCATIONS:
Overall Officials: François Luthi, MD, Principal Investigator — Clinique Romande de Readaptation
Locations (1):
- Clinique Romande de Readaptation, Sion, Valais, Switzerland

REFERENCES:
- [Derived] Plomb-Holmes C, Hilfiker R, Leger B, Luthi F. Impact of a non-return-to-work prognostic model (WORRK) on allocation to rehabilitation clinical pathways: A single centre parallel group randomised trial. PLoS One. 2018 Aug 2;13(8):e0201687. doi: 10.1371/journal.pone.0201687. eCollection 2018. PMID 30071081